CLINICAL TRIAL: NCT07045064
Title: Aerobic Versus Resistive Intradialytic Training Effect on Atherogeinc Index in Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Rezk Asad Rasheed, lecturer assistant at faculty of physical therapy Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: exerciseinhemodialysispatients
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
MeSH Terms: interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- arm 1 intervintion : aerobic exercise training without medication (Experimental): Group A:twenty patients of both sex Iintervention :moderate intensity intradialytic aerobic training for 12 weeks. (3 times per week). Using Horizontal electromagnetically braked cycle ergometer during the first half of the dialysis session.
  (1) Frequency: received intradialytic, lower-limb, cycling exercise three times per week on alternative days (2) Intensity: the intensity of exercise will be at 12-14 based on the Borg's Perceived Exertion Rating Scale.(a rating of 6 perceiving "no exertion at all" to 20 perceiving a "maximal exertion" of effort) ,Appropriate speed and grade of resistance were adjusted to achieve the required intensity. (3) Time: each session consisted of a a 5-min warm-up in form of ankle pump exercises, 20-min moderate intensity exercise, and 5-min cool-down phase in form of ankle pump exercise.
  Interventions: Other: Aerobic exercise without medication
- arm2 intervinsion :resistive exercise training without medication (Experimental): Grob B Twenty patients of both sex intervention :this group will participate in moderate intensity intradialytic resistive training without medication for 12 weeks . (3 sessions per week) using ankle weights.
  During session: The warming up phase for 5-minute in form of ankle pump exercises, then the main exercise phase and then cooling down phase for 5 minutes. in form of ankle pump exercises.
  The training protocol consisted of five lower-body resistance exercises using ankle weights 3 days/week, The intensity of the program will be moderate, starting with two sets of each exercise at 60% of each patient's three repetition max (3-RM) strength, progressing to three sets per session, with additional weight added as tolerated.
  Interventions: Other: resistive exercise without medication
- arm3 intervention : circulatory exercises training without medication (Experimental): Group C this group will include 20 patients of both sex intervension : patients will participate in ankle pump exercises and will be evaluated at the beginning and at the end of the study.
  Interventions: Other: circulatory exercise without medication

INTERVENTIONS:
Other: Aerobic exercise without medication — twenty patients will participate in moderate intensity intradialytic aerobic training for 12 weeks. (3 times per week). Using Horizontal electromagnetically braked cycle ergometer during the first half of the dialysis session.
  (1) Frequency: received intradialytic, lower-limb, cycling exercise three times per week on alternative days (2) Intensity: the intensity of exercise will be at 12-14 (moderate-intensity: somewhat hard or reports of feeling a little bit tired but still ok to continue) based on the Borg's Perceived Exertion Rating Scale Appendix III (a rating of 6 perceiving "no exertion at all" to 20 perceiving a "maximal exertion" of effort) ,Appropriate speed and grade of resistance were adjusted to achieve the required intensity. (3) Time: the duration of each exercise session consisted of a 5-min warm-up in form of circulatory exercise.
  Arms: arm 1 intervintion : aerobic exercise training without medication
Other: resistive exercise without medication — Twenty patients will participate in moderate intensity intradialytic resistive training for 12 weeks. (3 sessions per week) using ankle weights.
  During session: The warming up phase for 5-minute in form of circulatory exercises, then the main exercise phase and then cooling down phase for 5 minutes. in form of circulatory exercises.
  The training protocol consisted of five lower-body resistance exercises using ankle weights 3 days/week, The intensity of the program will be moderate, starting with two sets of each exercise at 60% of each patient's three repetition max (3-RM) strength, progressing to three sets per session, with additional weight added as tolerated
  Arms: arm2 intervinsion :resistive exercise training without medication
Other: circulatory exercise without medication — this group will include 20 patients will participate in circulatory exercises and will be evaluated at the beginning and at the end of the study.
  Arms: arm3 intervention : circulatory exercises training without medication

SUMMARY:
the goal of the clinical trial is to study the effect of aerobic and resistive exercises on atherogenic index in hemodialysis patients the study will include three groups of both sex the first group will participate in aerobic exercise ,the second group will participate in resistive exercise and the third group will be control group

DETAILED DESCRIPTION:
This study will be carried out on sixty male and female patients. They will be recruited from National Institute of Kidney and Urology, Mataria,Their ages will be ranged from (40-60) years old these patients will be assigned into three groups (A, B and C). The design of this study will be a randomized controlled trail (RCT).The patients will be informed about the study procedure and signed the informed consent prepared for this study . The study will follow the instructions of ethical committee of faculty of physical therapy, Cairo University. Inclusive criteria

1. Maintenance hemodialysis ≥ 3 months.
2. BMI will be ranged from 18.5 to 29.9 kg/m².
3. Age ≥ 40years and ≤ 60 years.
4. Hemodialysis 3 times a week.

Exclusive criteria:

1. patients suffered from any central and peripheral nervous system diseases.
2. patients suffered from serious complications, such as heart failure, severe infection and malignant tumor.
3. uncontrolled hypertension with systolic blood pressure ⩾200 mm Hg and/or diastolic blood pressure ⩾120 mm Hg,
4. unstable angina

ELIGIBILITY:
Inclusion Criteria:

.Maintenance hemodialysis ≥ 3 months. .BMI will be ranged from 18.5 to 29.9 kg/m². .Age ≥ 40years and ≤ 60 years. .Hemodialysis 3 times a week.

Exclusion Criteria:

.patients suffered from any central and peripheral nervous system diseases. .patients suffered from serious complications, such as heart failure, severe infection and malignant tumor.

.uncontrolled hypertension with systolic blood pressure ⩾200 mm Hg and/or diastolic blood pressure ⩾120 mm Hg.

.unstable angina

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
atherogenic index | three months
  aterogenic index will be measured through blood test ,an AIP value of under 0.11 is associated with low risk of CVD; the values between 0.11 to 0.21 and upper than 0.21 are associated with intermediate and increased risks, respectively

CONTACTS AND LOCATIONS:
Overall Officials: nesreen Vice Dean faculty of physical therapy, Professor, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - National Institute of Kidney and Urology, Mataria, Cairo, Select State
  - National Institute of Kidney and Urology, Mataria, Cairo

IPD SHARING:
Plan to Share IPD: No